CLINICAL TRIAL: NCT01252927
Title: Evaluation of a Gatekeeper Training Program as Suicide Intervention Training for Medical Students
Brief Title: Evaluation of a Gatekeeper Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Principal Investigator, Shay-Lee Bolton, PhD, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H2009:073
Record Dates: First submitted 2010-08-18; First posted 2010-12-03 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASIST intervention (Experimental): The gatekeeper training intervention group received the Applied Suicide Intervention Skills Training (ASIST) 10.0 in addition to TAU. ASIST is a two-day (fourteen hour), intensive, interactive and practice-dominated course aimed at enabling people to recognize risk and learn how to intervene immediately to prevent suicide. The intervention was offered to students on a weekend and was conducted by three senior ASIST trainers and one junior trainer, with two trainers assigned to each training group.
  Interventions: Other: ASIST
- Control group: training as usual (No Intervention): Training as usual consisted of didactic teaching and a tutorial with case-based examples around suicide risk factors in their first year of medical school. Third- and fourth-year students may also have the opportunity to practice their skills with real patients during their clerkship rotations or in the emergency department.

INTERVENTIONS:
Other: ASIST — The gatekeeper training intervention group will receive the Applied Suicide Intervention Skills Training (ASIST) workshop in addition to training as usual. ASIST is a 2-day intensive, interactive and practice-dominated course aimed at enabling people to recognize risk and learn how to intervene immediately to prevent suicide.
  Arms: ASIST intervention

SUMMARY:
The main objective of the proposed study is to evaluate the efficacy of a gatekeeper training suicide intervention program, Applied Suicide Intervention Skills Training (ASIST), in improving medical students' knowledge about suicide intervention, impact of attitudes on someone at risk for suicide and competent use of intervention skills to recognize risk and intervene effectively compared to medical education as usual. This research project will be undertaken using a randomized-controlled trial design. Questionnaires and objective structured clinical examinations using simulated patients will be completed at three time points: 1) before training, 2) after training, and 3) at one year following the training. Medical students' clinical skills in recognizing risk and intervening with simulated patients, as well as knowledge about suicide intervention and the impact of attitudes on someone at risk for suicide will be evaluated.

DETAILED DESCRIPTION:
The current proposal plans to implement and evaluate a secondary suicide intervention skills training program (gatekeeper training) in medical school students in Winnipeg, Manitoba, Canada. The main objective of the current proposal is to evaluate the effectiveness of a gatekeeper training program, Applied Suicide Intervention Skills Training (ASIST), in improving medical students' intervention skills with suicidal patients compared to training as usual. Secondary aims include comparisons of changes in knowledge, perceived competence and attitudes around suicide.

Findings from previous studies have demonstrated a significant positive effect of gatekeeper training on suicide prevention attitudes, skills and knowledge. As well, general studies in medical education reveal that students who have been able to practice, observe, and receive feedback in small groups showed an improvement in skills and confidence over those who were given didactic teaching only. Therefore, the investigators anticipate that the ASIST training program will significantly improve medical students' knowledge about suicide intervention, and will increase their recognition and response to suicide risk compared to education as usual. The investigators also expect that ASIST training will help them to understand the impact of attitudes on suicide prevention, and will increase their perceived competence and ability to recognize and treat a suicidal individual compare over training as usual. It is hypothesized that medical students trained in ASIST will differ significantly in their ability to correctly recognize and intervene with suicidal individuals based on their use of a standardized suicide intervention model and objective assessment using standardized patients.

ELIGIBILITY:
Inclusion Criteria:

* all medical students at University of Manitoba

Exclusion Criteria:

* those who choose not to participate
* those who have already taken ASIST training or related SafeTALK training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2011-03-27 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-08-01 (Actual)

PRIMARY OUTCOMES:
OSCE checklist total score | 1 week before training, 1 week following training, and 4 years following training
  Four Objective Structured Clinical Examinations (OSCEs) stations were developed for each time point in the study. All student-patient interactions were videotaped. Raters blind to the student's group assignment rated the videos according to a checklist of desired gatekeeper behaviors based on the key components of the ASIST program. A total score was the sum of all behaviours performed.
SIRI-2 score | 1 week before training, 1 week following training, and 4 years following training
  The Suicide Intervention Response Inventory (SIRI-2) is a self-administered questionnaire designed to measure competence in choosing appropriate responses to a series of clinical scenarios with suicidal individuals. It contains 25 items, each of which consists of a "client" remark and two "helper" responses. Respondents were instructed to evaluate the appropriateness of each of the two helper responses on a 7-point Likert scale, ranging from +3 (highly appropriate response) through 0 (neither appropriate nor inappropriate response) to -3 (highly inappropriate response). Ratings by a group of expert suicidologists and crisis interventionists provided a mean expert response criterion against which individual respondents are compared. The sum of the absolute value of the differences between the students' rating and the mean response from experts was calculated to obtain an overall score of how well the student performed with respect to expert responses.
OSCE global rating total score | 1 week before training, 1 week following training, and 4 years following training
  Four Objective Structured Clinical Examinations (OSCEs) stations were developed for each time point in the study. All student-patient interactions were videotaped. Raters blind to the student's group assignment rated the videos. Raters were asked to give a global rating score according to the performance of each student in each of the 3 key areas trained by the ASIST program, and a global rating of the student's performance on the station in general. The sum of all global ratings was used to determine a total score.

SECONDARY OUTCOMES:
self-perceived knowledge about suicide | 1 week before training, 1 week following training, and 4 years following training
  A single question measured the level of knowledge about suicide that the individual believes they have. Response options were on a 4-point Likert scale from very to not at all.
self-perceived skill in helping a suicidal individual | 1 week before training, 1 week following training, and 4 years following training
  A single question measured the level of ability that the individual believes they have in helping a suicidal person. Response options were on a 4-point Likert scale from very to not at all.
self-perceived confidence in helping a suicidal individual | 1 week before training, 1 week following training, and 4 years following training
  A single question measured the level of confidence that the individual believes they have in helping a suicidal person. Response options were on a 4-point Likert scale from very to not at all.
Attitudes towards suicide total score | 1 week before training, 1 week following training, and 4 years following training
  The Attitudes Towards Suicide Questionnaire (ATTS) was used to measure attitudes toward suicide. This scale is comprised of 37 items. Each item is rated on a 5-point Likert scale ranging from Strongly Disagree (1) to Strongly Agree (5). The total score of all 37 items was used for evaluation.
self-perceived preparedness | 1 week before training, 1 week following training, and 4 years following training
  A single question measured the level of preparedness that the individual believes they have in dealing with a suicidal individual. Response options were on a 4-point Likert scale from very to not at all.
Total score on Interpersonal Skills Rating Scale | 1 week before training, 1 week following training, and 4 years following training
  Interpersonal skills as rated by standardized patients in the OSCE setting according to the Interpersonal Skills Rating Scale. The IPS Rating Scale used 13 items to evaluate communication skills in the OSCE setting between patient and student from the patient's perspective, and included concepts such as empathy, respect, sensitivity, and listening skills. Each item was scored on a 7-point Likert scale from strongly agree to strongly disagree. The sum score of all 13 items was used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shay-Lee Bolton, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada